CLINICAL TRIAL: NCT05841823
Title: The Efficacy of Virtual Reality Exposure Therapy for the Treatment of Alcohol Use Disorder Among Adult Males: A Randomized Controlled Trial Comparing With Acceptance and Commitment Therapy and Treatment-as-usual
Brief Title: Virtual Reality Exposure Therapy in the Treatment of Alcohol Use Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Henan Medical University (Other)
Responsible Party: Principal Investigator, Mohammad Farris Iman Leong Bin Abdullah, Dr., Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XYEFYLL-(Research)-2022-29
Record Dates: First submitted 2023-04-06; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Alcohol Use Disorder
Keywords: alcohol use disorder; acceptance and commitment therapy; virtual reality exposure therapy; randomized controlled trial
MeSH Terms: conditions — Alcoholism | interventions — Virtual Reality Exposure Therapy; Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: multicenter, three-armed, parallel, single blind randomized control trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The allocation sequence is concealed in opaque, sequential numbered envelope. The randomization will be carried out by the research assistant which is not involved in the study. The data collection will also be carried out by the research assistant who did not know about the objective of the study. Hence, this is a three-armed parallel group single blind randomized controlled trial. The subjects are not blinded as they would have known which intervention they are in as the intervention procedures are different.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality exposure therapy (VRET) (Experimental): In this group, each session of VRET will last 25 minutes and consists of three parts: 5 minutes of relaxation, 10 minutes of exposure to high-risk situation and 10 minutes of exposure to aversive situation. Each participants will receive 20 sessions of VRET, 5 sessions per week for 4 weeks.
  Interventions: Behavioral: Virtual reality exposure therapy (VRET)
- Acceptance and commitment therapy (ACT) (Active Comparator): In this group, participants will receive a 50-minutes ACT session per week for 4 weeks. Hence, a total of 4 sessions will be administered to each participant.
  Interventions: Behavioral: Acceptance and commitment therapy (ACT)
- Treatment-as-usual control (TAU) (No Intervention): While for the control group, participants will receive non-specific ingredients of the psychotherapeutic approach schedule at a 50-minutes session per week for 4 weeks.

INTERVENTIONS:
Behavioral: Virtual reality exposure therapy (VRET) — The relaxation scene includes four beautiful landscapes, and patients can choose any of these four, as perceived to be the most comfortable landscape. The visual stimulation of high-risk scene is designed as any combination of four different scenes (street barbecue stands, restaurant, bar and home) and four kinds of alcoholic beverages (Chinese liquor, beer, grape wine and cocktail), which are customized according to the patient's personal preference. At the same time, the odor of the alcoholic beverage of the patient's choice will be provided as an olfactory stimulation. The aversive situation will be the visual and auditory stimulation provided by a video of an alcoholic vomiting, while olfactory stimulation will be provided by cotton balls soaked in fermented dairy products.
  Arms: Virtual reality exposure therapy (VRET)
Behavioral: Acceptance and commitment therapy (ACT) — The initial session began with case formulation. Subsequent sessions involved learning on acceptance and acknowledgement of unpleasant thoughts and feelings associated with alcohol craving and clinical features of alcohol use disorder, cognitive defusion on how to dissociate self avoidance of unpleasant thoughts and feelings, learning and practicing mindfulness exercise (such as mindfulness breathing) to make self aware of the many things that occurred presently which can be enjoyed and focus on rather than focusing on unpleasant thoughts and feelings, and learning to be aware of the safe self which is separated from the unpleasant thoughts and feelings and identifying values in life and strategies to achieve these values (therapeutic processes in hexaflex).
  Arms: Acceptance and commitment therapy (ACT)

SUMMARY:
This study aims to compare the efficacy of two types of interventions, which are acceptance and commitment therapy (ACT) as compared with virtual reality exposure therapy (VRET) for alleviating psychological dependence on alcohol and preventing relapse. It also assesses the changes of EEG in patients with alcohol use disorder after completion of the above related interventions.

In this study 120 subjects with alcohol use disorder who have completed 2 weeks of in-patient detoxification will be randomized into three groups (VRET, ACT and treatment-as-usual control groups) and undergo respective interventions. Then assessment will be performed at four timelines (baseline, 4 weeks after baseline which is immediately after completion of intervention, 12 weeks after baseline, and 24 weeks after baseline assessment).

DETAILED DESCRIPTION:
The approval of the study was obtained from the Human Research Ethics Committee of Xinxiang Medical University and from the Human Research Ethics Committee of Universiti Sains Malaysia. The study will be conducted according to the Declaration of Helsinki 1974 and its subsequent amendments and abide by the Good Clinical Practice Guidelines for Clinical Trial in Malaysia. If there is any amendments, for example in the eligibility criteria, study population, study procedures, interventions, data collection, data analysis; it will be informed in writing to the Human Research Ethics Committee of Xinxiang Medical University and the Human Research Ethics Committee of Universiti Sains Malaysia.

Prior to participation in the trial, participants will be informed of their right to withdraw from the trial at any time and the data collected will be discarded immediately and will not be used for the study. Participants will be reminded that all personal identifiable information will not be used and only group data will be analyzed and published. They will be assured of their anonymity for participating in the trial. The participants will be assured that the data collected will only be used for research purposes and the findings will not be recorded in their case files. All participants will be assigned a research number for identification purposes, for example "VT 001". All the data collected from the participants will be stored in the research file which will be locked in a file cabinet, whereby the key will be kept by the principal investigator. Data collected may also be stored in thumb drive and lap top which is only accessible by the research team and the principal investigator. Prior to participation, all the participants will also be informed regarding the study purposes, study procedures, and the risks and benefits of participating in the study. The findings of the study will be published in academic journals and presented in conferences or symposia. As for publication of research findings in academic journals, the principal investigator will be the corresponding author while the other authorship will be determined according to the the International Committee of Medical Journal Editors' recommendations. All the investigators in the research team declared that there is no competing interest in term of financial gain or the conduct of this study.

Participants who experienced any adverse effects (AE) will be withdrawn from the study. AE is any untoward medical events which occurred with or without causal relationship with the study's intervention. In order to monitor AE during the trial, all participants will be given a trial card which contains the name, contact number and email of the members of the research team. They are encouraged to contact the research team member in charge if there is any occurrence of AE. The occurrence of AE will then be reported to the "adverse effect" section of the trial's case report form. The details of the AE reporting will contain information, such as the name of the AE, the date of occurrence and date of resolution, severity, AE relationship with the study intervention, treatment of AE, and the outcome (resolve or still on-going). The AE which may lead to withdrawal of participants from the trial are: (1) adverse reaction which is not related to the study intervention but cause discomfort to the participants, (2) adverse reaction which is related to the study intervention (probiotic, ACT and/or placebo), and (3) any changes in behavior, temperament, personality, psychotic symptoms, and suicidal tendency that occurred after the study intervention began (VRET, ACT or TAU). All AE should be reported to the Human Research Ethics Committee of Xinxiang Medical University and Universiti Sains Malaysia and investigation should be carried out. If there is any safety concerns regarding the administration of the study intervention (VRET, ACT, and TAU), such as deliberate self-harm, suicidal tendency, bacterial infection, sepsis, hospitalization due to psychological adverse effect arise from the intervention, or mortality; there it is an indication for premature termination of the trial after an interim analysis.

The principal investigator will lead the trial center and will coordinate closely with the research and site coordinators in a day-to-day basis involving in the conduct of the clinical trial, subject recruitment, and data collection. A trial monitoring unit will also be set up which will be chaired by the principal investigator, whereby weekly meeting will be held to discuss on the conduct of the trial, auditing of the trial, and prepare report to be submitted to the Human Ethics Committee of Xinxiang Medical University and Universiti Sains Malaysia. The monitoring of trial data and auditing of the trial will be managed by the clinical trial coordination unit of the 2nd Affiliated Hospital of Xinxiang Medical University and Advanced Medical and Dental Institute, Universiti Sains Malaysia, which are independent of the funder. Interim analysis will be carried out if there is such necessity for premature termination of the trial based on assessment and auditing of the trial data.

The estimated sample size will be calculated using the G*Power 3.1.9.7 sample size calculator using the sample size calculation for repeated measure ANOVA, within-between interaction, whereby the type I error was 0.05, the power was 0.8, the number of groups was three, the number of measures was four, and the effect size was 0.14. The estimated total sample size needed was 120 (after inclusion of 30% drop out), in which 40 subjects per group is required.

Initially, all subjects enrolled in the study will receive 2 weeks of conventional treatment for AD which includes benzodiazepine (BZD) replacement therapy for detoxification, low-dose antipsychotics, adequate vitamin B12 dosage and supportive treatment for symptomatic relief. The conventional treatment is administered to ensure that all the subjects who participated in this study will have stopped drinking for two weeks before the start of the study, and their physical withdrawal symptoms will be relived after two-week medication, mainly BZD replacement therapy.

Then, all subjects will be randomly assigned to three groups: i) patients provided with ACT for 4 weeks in combination with conventional treatment, ii) provided with VRET for 4 weeks in combination with conventional treatment, and iii) patients receiving only conventional treatment and non-specific ingredients of the psychotherapeutic approach for 4 weeks.

The ACT intervention will be conducted individually for each session. The ACT modules cover 4 sessions, 1 hour in each session. The sessions will be held once a week. The VRET intervention will be conducted in a single patient for each session. The total course of VRET includes 20 sessions, 25 minutes in each session. The sessions will be held five times a week, hence a total duration of 4 weeks needed.

While for the control group, they will receive non-specific ingredients of the psychotherapeutic approach, such as psychological understanding to the management of an individual patient, identifying current problems, providing opportunities for disclosure, and reassurance. They will be given equal amount of time and attention from the professional figure compared to the intervention groups, whereby they will also attach to a 4-session programme (with one session per week for total duration of 4 weeks). After completing the study (after t3 assessment), they will be offered for either ACT or VRET for treatment.

Assessments will be performed across four timelines: pre-intervention (baseline- the second weekend after admission), 4 weeks after baseline (immediately after completion of intervention), 12 weeks after baseline (follow-up after discharge), and 24 weeks after baseline (follow-up after discharge).

At each assessment timepoints, the subjects will undergo the assessments which include the following:

1. For assessment of the degree of severity of alcohol use disorder related symptoms, several clinical questionnaire tools will be used such as i) Alcohol Use Disorders Identification Test (AUDIT), ii) Clinical Institute Withdrawal Assessment-Alcohol, Revised (CIWA-Ar), and iii) Penn Alcohol Craving Scale (PACS). All questionnaires will be administered by clinicians.
2. For exploration of the objective indicators related to the severity of alcohol craving, ERP evoked by alcohol cue reactivity will be detected.
3. For assessment of the emotional aspects of patients with AD, several emotional rating scales will be used such as i) Hamilton Anxiety Scale (HAMA), and ii) Hamilton Depression Scale (HAMD).

All data analysis will be performed using SPSS software version 25.0 (SPSS Inc, Chicago, IL, USA). Descriptive statistics for socio-demographic and clinical characteristics, CIWA-Ar, PACS, AUDIT, VAS, HAMD, and HAMA scores, ERP analysis, and serum electrolytes, liver function test, and γ-glutamyl transpeptidase levels will be computed. All categorical variables will be presented in frequency and percentage, while all continuous variables will be reported in mean and standard deviation or median and interquartile range, depending on normality. While differences in the CIWA-Ar, PACS, AUDIT, HAMD, and HAMA scores, and ERP analysis between groups at the same time point will be assessed suing one way ANOVA. Finally, the differences in the CIWA-Ar, PACS, AUDIT, VAS, HAMD, and HAMA scores, and ERP analysis between groups and within group at different time points will be evaluated using two-way repeated measure ANOVA. Statistical significance was set at p < 0.05 and two-sided.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized patients diagnosed with alcohol use disorder (confirmed by the relevant diagnostic criteria of Diagnostic and Statistical Manual of Mental Disorders-V).
2. Male, age 18 to 55 years old, Han nationality, junior high school education or above, right-handed (because of the difference in EEG between right-hand and left-hand).
3. Those with normal eyesight (including corrected vision).

Exclusion Criteria:

1. Those with current and lifetime history of abuse of any other psychoactive substances (except tobacco).
2. Those with current and lifetime history of other mental diseases.
3. Those with current and lifetime history of central nervous system diseases or serious physical illnesses.
4. Those who are unable to complete the EEG detection or psychological scale assessment.
5. Those who are unable to cooperate with ACT or VRET, or who are seriously uncomfortable with psychotherapy.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only male subjects are recruited
Enrollment: 120 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Alcohol Use Disorders Identification Test (AUDIT) score across four timelines | At four time points of assessment: t0 (baseline) = before starting intervention, t1 = 4 weeks which is immediately after completion of intervention, t2 = 12 weeks after intervention began, and t3 = 24 weeks after intervention began
  This questionnaire can differentiate drinkers from mild to severe. The scale consists of 10 questions, of which three relate to the amount and frequency of alcohol consumption, three relate to alcohol dependence and four involve in various problems caused by alcohol. The score of the scale ≥ 8 is positive. In general, those with high scores on the first three questions but low scores on the rest suggest serious harmful drinking; High scores in questions 4, 5 and 6 indicate alcohol dependence; High scores in the final section indicate that drinking has caused harm. The reliability and validity of the Chinese version are 0.782. Factor analysis showed that indeed the Chinese version of the AUDIT comprised of three factors and had good convergent and discriminant validity. Total score ranged from 0 to 40.
Change in Clinical Institute Withdrawal Assessment-Alcohol, Revised (CIWA-Ar) score across four timelines | At four time points of assessment: t0 (baseline) = before starting intervention, t1 = 4 weeks which is immediately after completion of intervention, t2 = 12 weeks after intervention began, and t3 = 24 weeks after intervention began
  The scale is a standard tool for quantifying the severity of alcohol withdrawal symptoms. The total score < 10 suggests mild withdrawal reaction. The score of 10 to 20 indicates moderate. The total score of more than 20 is considered severe. A severe total score is associated with a risk of delirium tremens and seizures. The reliability of the Chinese version of CIWA-Ar was good with Cronbach's α of 0.83. Total score ranged from 0 to 30.
Change in Penn Alcohol Craving Scale (PACS) score across four timelines | At four time points of assessment: t0 (baseline) = before starting intervention, t1 = 4 weeks which is immediately after completion of intervention, t2 = 12 weeks after intervention began, and t3 = 24 weeks after intervention began
  This questionnaire consists of five items to evaluate the severity of craving, including frequency, intensity, duration, difficulty of coping, and average craving degree. It is a seven-point scale from 0 to 6, with 0 being none and 6 being extremely severe. The subjects will be asked to answer questions according to the situation in the past week. The reliability of the Chinese version of PACS was good at Cronbach's α of 0.97. Total score ranged from 0 to 30.

SECONDARY OUTCOMES:
Change in Hamilton Anxiety Rating Scale (HAM-A) score across four timelines | At four time points of assessment: t0 (baseline) = before starting intervention, t1 = 4 weeks which is immediately after completion of intervention, t2 = 12 weeks after intervention began, and t3 = 24 weeks after intervention began
  The HAM-A is an observer administered instrument to assess the severity of anxiety symptoms. It consists of 14 items which assess 14 anxiety symptoms. Each item is scored in a Likert scale ranging from 0 (not present) to 4 (severe). A total score of < 17 indicates mild severity, 18 to 24 denotes mild to moderate, 25 to 30 indicates moderate to severe, and > 30 indicates severe. The instrument has been translated and validated in the Chinese population with an excellent internal consistency with Cronbach's α of 0.93. Total score ranged from 0 to 56.
Change in Hamilton Depression Rating Scale (HAM-D) score across four timelines | At four time points of assessment: t0 (baseline) = before starting intervention, t1 = 4 weeks which is immediately after completion of intervention, t2 = 12 weeks after intervention began, and t3 = 24 weeks after intervention began
  The HAM-D is an observer administered instrument to assess the severity of depressive symptoms. The HAM-D consists of 21 items, but is scored on the first 17 items. The higher the score, the greater is the severity of depressive symptoms. The interpretation of the total score are such that, score of 0 to 7 indicates normal, 8 to 16 denotes mild depression, 17 to 23 indicates moderate depression, and 24 and above denotes severe depression. The instrument was translated and validated in the Chinese population with an acceptable internal consistency with Cronbach's α of 0.714. Total score ranged from 0 to 77.

OTHER OUTCOMES:
Change in event-related potential (ERP) in EEG across four timelines | At four time points of assessment: t0 (baseline) = before starting intervention, t1 = 4 weeks which is immediately after completion of intervention, t2 = 12 weeks after intervention began, and t3 = 24 weeks after intervention began
  Visual stimuli will be presented by the E-Prime 2.0 software. There are three types of visual stimuli, such as (a) images related to alcohol cues (for example common places where alcohol is consumed, habitual alcohol products, people drinking alcohol, etc.), (b) neutral images which are not related to alcohol cues, and (c) task-related images which require key operation. The EEG monitoring and recording will be carried out while the participants watch the stimulation paradigm. EEG signal monitoring and recording is performed using the Brain Amp MR-32 instrument and through the Brian Vision Recorder software.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Farris Iman Leong Bin Abdullah, Dr Psych, Principal Investigator — Advanced Medical and Dental Institute, Universiti Sains Malaysia (USM)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deng H, Zhang R, Wang C, Zhang B, Wang J, Wang S, Zhang J, Shari NI, Leong Bin Abdullah MFI. The efficacy of virtual reality exposure therapy for the treatment of alcohol use disorder among adult males: a randomized controlled trial comparing with acceptance and commitment therapy and treatment as usual. Front Psychiatry. 2023 Aug 22;14:1215963. doi: 10.3389/fpsyt.2023.1215963. eCollection 2023. PMID 37674551